CLINICAL TRIAL: NCT02165592
Title: Assessment and Identification of Proprioceptive and Functional Changes in Patients With Hemophilia of the Region of Murcia.
Brief Title: Assessment of Proprioceptive and Functional Characteristics in Patients With Hemophilia
Acronym: HE-BALANCE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, RUBÉN CUESTA-BARRIUSO, PhD, Universidad Católica San Antonio de Murcia
Other Study IDs: UCAM-2; UCAM-2
Record Dates: First submitted 2014-06-13; First posted 2014-06-17 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-09

CONDITIONS: Hemophilia
Keywords: Hemophilia; Arthropathy; Range of Motion; Strength; Proprioception; Gait; Quality of Life
MeSH Terms: conditions — Hemophilia A; Joint Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with hemophilia: Patients with hemophilia who meet the inclusion criteria

SUMMARY:
Analyze and evaluate the skeletal muscle of patients affected with hemophilia in the Region of Murcia.

* Describe the periarticular muscular deficit of the lower limbs, depending on the degree of injury: acute and chronic, or subacute.
* Identify the range of motion of joints with higher prevalence of hemophilic arthropathy.
* Detect the biomechanical changes of the lower limbs and their impact on gait in patients with hemophilia.
* Assess the factors that influence the perception of illness and quality of life of patients with hemophilia.

DETAILED DESCRIPTION:
Descriptive study of joint involvement in hemophilia patients with and without a history of hemarthrosis in lower limbs.

Descriptive study of alterations in the strength of the periarticular muscles of lower limbs as a result of acute conditions or the development of chronic articular sequelae.

Descriptive study of the biomechanical alterations in weight-bearing joints of lower limbs and their impact on gait in patients with hemophilia.

Descriptive study of the relationship between skeletal muscle pathology in patients with hemophilia and their perceptions of it and their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hemophilia A and B
* Patients of all ages (from 6 to 70 years).
* With or without joint damage clinically diagnosed, and with or without a previous history of hemarthrosis joint load legs.
* Residents in the Autonomous Community of the Region of Murcia.

Exclusion Criteria:

* Patients without ambulation
* Patients diagnosed with other congenital coagulopathy (von Willebrand disease, etc..).
* Patients with neurological or cognitive impairments that prevent understanding the questionnaires and physical tests.

Ages: 6 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients from the Murcia Regional Hemophilia Association
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2015-09; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Assess the range of motion | Screening visit
  Assess the range of motion of elbow, knee and ankle (using a goniometric evaluation).
Assess the muscular strength | Screening visit
  Assess the muscular strength of arm, thigh and leg (through measurement of muscle balance).
Assess the joint pain | Screening visit
  Joint pain (VAS scale with the use of a pressure algometer).
Assess the variables of strength | Screening visit
  Assessment of variables of vertical strength, medio-lateral and anterior-posterior in jump and incorporation from the sitting position.
Assess the peak force | Screening visit
  Functional assessment of peak force, force production per unit time and subsequent stabilization in standing (in jump and in the passage from the sitting position to standing position, respectively, using a force platform).
Assess the contractile activity | Screening visit
  Assessment of miotendinous contractile activity in the patellar tendon and Achilles, in jump (CMJ-stiffness test).
Assess the state joint | Screening visit
  State joint (applying Hemophilia Joint Health Score questionnaire).
Assess the list of activities | Screening visit
  List of activities in hemophilia (completing the autocuestionario Hemophilia Activities List).
Assess the physical performance | Screening visit
  Perception of physical performance (with the HEP-Test-Q questionnaire)
Assess the health Profile | Screening visit
  Health Profile (using the scale Nottingham health profile)
Assess the quality of life | Screening visit
  Quality of life (using the SF-36 and Haemo-QoL-36 questionnaire).

SECONDARY OUTCOMES:
Age, sex, weight of the patients with hemophilia | Screening visit
Diagnosis, severity of hemophilia, type of treatment (prophylactic or on-demand) and inhibitors | Screening visit
Frequency of joint bleeds in the previous month and bleeding during the assessment | Screening visit

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Católica San Antonio, Murcia, Murcia, Murcia, Spain